CLINICAL TRIAL: NCT01431560
Title: Outcomes of Operative Treatment of Unstable Ankle Fracture - Comparison Between Metallic and Biodegradable Implants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Police Hospital (Other Government)
Responsible Party: Principal Investigator, Jung Ho Noh, Orthopaedic Surgeon, National Police Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: National Police Hospital
Record Dates: First submitted 2011-09-02; First posted 2011-09-09 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Ankle Fracture
Keywords: ankle; metallic; biodegradable; Freedom
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metallic implant (Active Comparator): fixation of the ankle fracture with metallic implants
  Interventions: Device: fixation of the ankle fracture (Solco )
- biodegradable implant (Active Comparator): fixation of the ankle fracture with Freedom plate and screws
  Interventions: Device: fixation of the ankle fracture (Freedom)

INTERVENTIONS:
Device: fixation of the ankle fracture (Solco ) — fixation with metallic implant
  Other Names: metallic implant: Solco
  Arms: metallic implant
Device: fixation of the ankle fracture (Freedom) — fixation with biodegradable implant
  Other Names: biodegradable implant: Freedom
  Arms: biodegradable implant

SUMMARY:
The purposes of this study are to compare the outcomes of the biodegradable implants for the fixation of ankle fracture and those of metallic implants, and to assess the problems of the biodegradable implants. Null hypothesis is that the clinical outcomes of biodegradable plate and screws for ankle fracture are not different from those of metallic implants.

ELIGIBILITY:
Inclusion Criteria:

* skeletally mature subjects (≥16 years old) with unilateral ankle fractures

Exclusion Criteria:

* subjects less than 16 years old,
* subjects not followed up at this hospital,
* multiple injuries,
* bilateral ankle fractures,
* open fractures,
* pathologic fractures,
* concomitant tibial shaft fractures,
* previous history of immobilization due to significant injury or a fracture of either ankle,
* significant peripheral neuropathy,
* soft tissue infection in the region on either injured ankle,
* or inability to complete the study protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
American Orthopaedic Foot and Ankle Society(AOFAS) score | 3 months, 6 months, 1 year
  change from baseline(3 months after surgery)

SECONDARY OUTCOMES:
Short Musculoskeletal Functional Assessment(SMFA) scale | 3 months, 6 months, 1 year
  change from baseline (3 months after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Jung Ho Noh, M.D., Ph.D., Principal Investigator — National Police Hospital, Korea, Republic of
Locations (1):
- National Police Hospital, Seoul, South Korea